CLINICAL TRIAL: NCT00182403
Title: Fixed Dose Unfractionated Heparin for Initial Treatment of Venous Thromboembolism
Brief Title: Fixed Dose Heparin Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMG-2005-FIDO; #NA3640
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Unfractionated Heparin; Low Molecular Weight Heparin; Venous Thromboembolism; APTT; Treatment
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: UFH 250 U/kg or LMWH 100 U/kg sc twice daily

SUMMARY:
FIDO was a multicentred randomized, open-label trial that compared fixed-dose UFH with fixed-dose LMWH for initial treatment of VTE. Patients were followed for 3 months during which they received warfarin (target INR 2.0-3.0).

DETAILED DESCRIPTION:
The general objective was to simplify and reduce the cost of treatment of acute venous thromboembolism (VTE).Specific objectives were to compare the efficacy, safety and cost effectiveness of unfractionated heparin (UFH) and low molecular weight heparin (LMWH) when each is administered subcutaneously (sc), twice daily, in weight -adjusted, fixed doses; and to determine if the anticoagulant response (anti-Factor Xa heparin levels, APTT results) influence efficacy and safety of UFH and LMWH, independently of dose.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of acute venous thromboembolism (VTE,DVT and /or PE)

Exclusion Criteria:

* Contraindication to subcutaneous (sc) route of administration (eg:shock (evidence of poor peripheral perfusion), major surgery within 48 hours)
* Active Bleeding process
* Comorbid condition limiting expected survival to less than 3 months
* Current treatment with therapeutic dose of UFH, LMWH, danaparoid sodium, or a direct thrombin inhibitor for more than 48 hours
* Currently on long term warfarin or heparin therapy
* Allergy to heparin or history of heparin induced thrombocytopenia
* Currently pregnant
* Contraindication to contrast media (eg: allergy or creatinine >200 umol/L).
* Currently enrolled or will be enrolled in a competing study
* Geographically inaccessible for follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866
Dates: Start 1998-09; Study Completion 2004-05

PRIMARY OUTCOMES:
Symptomatic Venous Thromboembolism
Major Bleeding
Death

SECONDARY OUTCOMES:
aXa ~6h after sc injection on 3rd day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MB Ph.D, Principal Investigator — Hamiton Health Sciences; Jim Julian, MMath, Principal Investigator — McMaster-Dept. of Clinical Epidemiology &Biostatistics
Locations (8):
- Canada (6):
  - Hamilton Health Sciences-General Campus, Hamilton, Ontario
  - Hamlton Health Sciences -McMaster Campus, Hamilton, Ontario
  - St. Joseph's Healthcare Centre, Hamilton, Ontario
  - Hamilton Health Sciences-Henderson Campus, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHA Pavillon du Saint-Sacrement, Québec, Quebec
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Middlemore, Otahuhu

REFERENCES:
- [Result] Kearon C, Ginsberg JS, Julian JA, Douketis J, Solymoss S, Ockelford P, Jackson S, Turpie AG, MacKinnon B, Hirsh J, Gent M; Fixed-Dose Heparin (FIDO) Investigators. Comparison of fixed-dose weight-adjusted unfractionated heparin and low-molecular-weight heparin for acute treatment of venous thromboembolism. JAMA. 2006 Aug 23;296(8):935-42. doi: 10.1001/jama.296.8.935. PMID 16926353